CLINICAL TRIAL: NCT06355453
Title: Evaluation of the Goldcrest Patch Performance
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-090-MIC-GES
Record Dates: First submitted 2024-03-11; First posted 2024-04-09 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Fetal Monitoring
Keywords: Fetal Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pregnant Woman Arm: Subjects will have Goldcrest patch and three Novii electrodes will be placed on the subjects abdomen.
  Interventions: Device: Goldcrest Patch and Three Patch Coupons
- Non-Pregnant Woman Arm: Subjects will have Goldcrest patch and Novii Patch and electrodes will be placed on the subjects abdomen.
  Interventions: Device: Goldcrest Patch and Novii Patch

INTERVENTIONS:
Device: Goldcrest Patch and Three Patch Coupons — Goldcrest patch and three patch coupons will be placed on subject abdomen for 18 hours (+/- 2 hours) of wear. Evaluation of skin integrity and patch performance will be assessed.
  Groups: Pregnant Woman Arm
Device: Goldcrest Patch and Novii Patch — Goldcrest patch and Novii patch will be placed on subject abdomen for 18 hours (+/- 2 hours) of wear. Evaluation of skin integrity and patch performance will be assessed.
  Groups: Non-Pregnant Woman Arm

SUMMARY:
The Novii Patch is an accessory to the Novii+ Pod that connects directly to the Novii+ Pod and contains the surface electrodes that attach to the abdomen.

The primary objective is to collect Data on Skin Integrity and Patch Adhesion Quality From the Patch After 18 Hours of Wear. The secondary objective is to evaluate fetal monitoring on adult pregnant females greater than 32 weeks gestation and non-pregnant females to collect data on electrical fetal, maternal, and uterine activity.

DETAILED DESCRIPTION:
The primary objective is to collect Data on Skin Integrity and Patch Adhesion Quality From the Patch After 18 Hours of Wear. The secondary objective is to evaluate fetal monitoring on adult pregnant females greater than 32 weeks gestation and non-pregnant females to collect data on electrical fetal, maternal, and uterine activity.

ELIGIBILITY:
Inclusion Criteria for all Subjects:

* Adult Females, 22 to 70 years of age.
* Must be able to read and speak English.
* Able and willing to provide written informed consent.

Inclusion criteria that apply to the pregnant person arm only:

- Pregnancy of greater than or equal to 32.0 weeks gestation per self-report.

Exclusion Criteria:

* Skin irregularities or other characteristic (such as scars, moles) on abdominal area that could interfere with completion of study procedures or identify a subject;
* Subjects who have implantable devices such as Transcutaneous Electrical Nerve Stimulation (TENS) machines, Cardiac Pacemakers or Cardiac Defibrillators
* Subjects expected to be at risk from participation for any reason, such as those with known allergy or sensitivity to adhesive materials that may be used in the study, such as silicone;
* Subjects over the age of 70;
* Unable to read or speak English language
* Direct employees or contractors of GE HealthCare, or any company that makes fetal monitoring devices.

Exclusion criteria that apply to specific arms only:

* Non-Pregnant Arm: Subjects who are currently pregnant, or unsure of pregnancy status per self-report;
* Pregnant Arm: Multiple gestation pregnancy or those self-reported to have been diagnosed as high risk by a provider (e.g., pre-eclampsia, gestational hypertension, being followed by a perinatologist).

Ages: 22 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Community sample in Milwaukee, Wisconsin area.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Collection of Skin Integrity Quality | 18 hours
  To collect of skin integrity quality from a skin assessment scale the from the patch's after 18-hours of wear.

SECONDARY OUTCOMES:
Collection of ECG Electrical Signal Data | 18 hours
  Collection of electrocardiogram (ECG) electrical signal data from the patch after 18 hours of wear.
Collection of Subject Activity | 18 hours
  Collect of subject activity data utilizing a subject questionnaire during the 18 hours of wear.
Collection of Patch Electrical Signal Data | 18 Hours
  Collection of electrical signal data from the patch's at the time of application for comparison to the electrical data after 18 hours of wear

OTHER OUTCOMES:
Safety Analysis | 4 months
  Analysis of adverse events will be listed per subject, summarized with counts and percentages of events, and summarized with counts and percentages of subjects with events.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Systems Engineering Manager, Principal Investigator — GE Healthcare
Locations (1):
- GE HealthCare Research Park, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
This is an early phase investigation of a device

REFERENCES:
- [Background] Lawrence A, Lewis L, Hofmeyr GJ, Dowswell T, Styles C. Maternal positions and mobility during first stage labour. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD003934. doi: 10.1002/14651858.CD003934.pub2. PMID 19370591
- [Background] McNichol L, Lund C, Rosen T, Gray M. Medical adhesives and patient safety: state of the science: consensus statements for the assessment, prevention, and treatment of adhesive-related skin injuries. Orthop Nurs. 2013 Sep-Oct;32(5):267-81. doi: 10.1097/NOR.0b013e3182a39caf. PMID 24022422